CLINICAL TRIAL: NCT00094783
Title: Real-Time MRI-Guided Percutaneous Intervention for Aorto-illac and Femoropopliteal, Artery Stenosis
Brief Title: MRI-Guided Balloon Angioplasty to Treat Blood Flow Blockage in the Legs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050007; 05-H-0007
Record Dates: First submitted 2004-10-22; First posted 2004-10-25 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-06-17

CONDITIONS: Cardiovascular Diseases
Keywords: Magnetic Resonance Imaging; Interventional MRI; Arterial Stenosis; Revascularization; Lllac Artery Stenosis; Peripheral Arterial Disease; Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases; Peripheral Arterial Disease

INTERVENTIONS:
Procedure: MRI

SUMMARY:
This study will examine the use of magnetic resonance imaging (MRI) instead of x-rays to guide angioplasty in patients who require these treatments to treat blockages in leg arteries. Angioplasty is a procedure in which a balloon is inflated in a blocked artery to improve blood flow. MRI uses a magnetic field and radio waves rather than x-rays to show pictures of body tissues and organs. MRI shows all soft tissue, including the arteries, blood, and other organs, while the usual x-ray technique shows only the lumen of the artery when it is filled with dye, but not the vessel walls.

Patients 18 years of age and older who require angioplasty with or without stenting to restore blood flow to the leg may be eligible for this study.

Participants undergo the usual angioplasty procedure. The skin in the patient's groin area is numbed and a catheter is placed into the groin artery. The patient is given a blood-thinning medicine, and then other catheters are inserted to measure blood pressure and to inject a contrast dye to take pictures. Balloon catheters are inflated to open the blockage and, if needed, stents are put in place to maintain the opening. When the blood thinner wears off, the catheters are removed.

Most of the procedure is conducted using MRI instead of X-rays to visualize the arteries and blockages. The patient is moved back and forth between the x-ray and MRI machines in a specially designed laboratory. If necessary, stenting, placement of a wire mesh to hold open the artery, is done using conventional x-ray techniques.

The entire procedure, including MRI, takes up to 4 hours.

DETAILED DESCRIPTION:
Cardiovascular interventional procedures are minimally-invasive, catheter-based treatments such as coronary artery angioplasty and stenting. These procedures generally can be conducted on awake patients with few complications, and were developed as alternatives to conventional open surgery. Conventional cardiovascular interventional procedures are conducted by physician manipulating medical devices inside patients under the guidance of fluoroscopic x-ray.

We have developed minimally-invasive cardiovascular interventional procedures using real-time magnetic resonance imaging. These procedures have the advantage of excellent imaging without surgery and without ionizing radiation exposure or toxic contrast agents (dyes). Moreover, because real time MRI can produce excellent images of soft tissue, blood, and of three-dimensional structures, it may be possible to guide minimally-invasive procedures not possible even with invasive surgery.

A state-of-the-art combined X-ray and MRI interventional suite has been constructed and equipped with real-time MRI image reconstruction for interventional experiments, patient monitoring and transport equipment for dual imaging modalities, and large-mammal preclinical simulation experiments. Preclinical experiments in a porcine model of surgical aortic coarctation have shown that real-time MRI guided percutaneous intervention can be conducted using entirely commercially-available devices approved by the US Food and Drug Administration.

The goal of this protocol is to test clinical peripheral artery revascularization procedures guided wholly-or in part by real-time MRI.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with known or suspected cardiovascular disease will be eligible for participation in this protocol. The patient is eligible under the following conditions:

* Patients age is greater than 18 years of age.
* Undergoing a clinically-indicated therapeutic peripheral artery catheterization procedure.
* Target peripheral artery is aorto-illac or femoropopliteal artery.
* Target peripheral artery stenoses, not occlusions, evident on magnetic resonance or x-ray angiography.

EXCLUSION CRITERIA:

Patients with absolute contraindications to MRI scanning will be excluded. These contraindications include patients with the following devices:

* Implanted cardiac pacemaker or defibrillator.
* Central nervous system aneurysm clips.
* Implanted neural stimulator.
* Cochlear implant.
* Ocular foreign body (e.g. metal shavings).
* Insulin pump.
* Metal shrapnel or bullet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2004-10-20; Study Completion 2008-06-17

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Guttman MA, Lederman RJ, Sorger JM, McVeigh ER. Real-time volume rendered MRI for interventional guidance. J Cardiovasc Magn Reson. 2002;4(4):431-42. doi: 10.1081/jcmr-120016382. PMID 12549231